CLINICAL TRIAL: NCT06494787
Title: A Phase 2 Study Using Aliya Pulsed Electric Field Ablation Plus Pembrolizumab for Sarcoma
Brief Title: A Phase 2 Study Using Aliya PEF Plus Pembro for Sarcoma
Acronym: SOC-2320
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Sarcoma Oncology Research Center, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOC-2320
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a phase 2 study to determine the efficacy and safety of the Aliya PEF System combined with pembrolizumab in treating patients with advanced soft tissue sarcoma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aliya PEF Plus Pembrolizumab (Experimental): This is an open label, phase 2 using Aliya PEF energy and Pembrolizumab 200 mg i.v. over 30 minutes every 3 weeks.
  Interventions: Combination Product: Aliya Pulse Electric Field sysem and pembrolizumab

INTERVENTIONS:
Combination Product: Aliya Pulse Electric Field sysem and pembrolizumab — This is a phase 2 study to determine the efficacy of the Aliya Pulse Electric Field system and pembrolizumab in prolonging progression free and overall survival of patients with advanced soft tissue sarcoma

SUMMARY:
The is a phase 2 that will evaluate the efficacy and safety of the Aliya PEF ablation system combined with pembrolizumab, an immune checkpoint inhibitor.in advanced soft tissue sarcoma. Twenty subjects will be treated.

DETAILED DESCRIPTION:
This is a Phase 2 study that will evaluate the efficacy and safety of the Aliya PEF ablation system plus pembrolizumab, an immune checkpoint inhibitor in advanced soft tissue sarcoma.

The AliyaTM System (Galvanize TherapeuticsTM) is a biphasic monopolar pulsed electric field (PEF) system that induces cell death in a manner independent of thermal processes, enabling focal ablation without denaturing stromal proteins or inducing significant muscle contraction. Pembrolizumab is a programmed death receptor-1 (PD-1)-blocking indicated for various malignancies including melanoma, non-small cell lung cancer, small cell lung cancer, head and neck squamous cell cancer, etc.Both Aliya and Pembrolizumab are FDA approved products.

Objectives:Primary: o evaluate progression free survival at 6 months; Secondary: To evaluate the objective response rate by RECIST v1.1 via CT scan or MRI at week 6 and every 6 weeks thereafter until end of treatment (EOT); to determine progression-free survival (PFS) at 6 months and overall survival, and to evaluate the incidence and grade of treatment related adverse events.

Exploratory: To evaluate PEF-Treated Dose-Response- Pre-PEF and follow-up as per standard of care after PEF energy delivery by RECIST v1.1 and iRECIST criteria, and to conduct biomarker analyses performed on tumor homogenate prep (THP) and lab blood draws collected at follow-up visits as per standard of care, which may include flow cytometry analyses of cell populations, cytokines, tumor-specific T-cell and B-cell populations, and tumor-specific IgG antibody quantities.The population to be studied include male and female subjects 18 years of age or older, of any ethnicity, with advanced soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ≥ 18 years of age
* Pathologically confirmed diagnosis of pleomorphic sarcoma, myxofibrosarcoma, leiomyosarcoma, liposarcoma, synovial sarcoma
* Previously treated or untreated patients
* Measurable disease with at least one target lesion amenable to PEF
* Life expectancy at least 3 months
* Adequate hematologic, liver and kidney function
* ECOG performance status of 0-1
* Willingness to sign informed consent
* Negative pregnancy test if female

Exclusion Criteria:

* Patients with untreated CNS disease
* Anticancer therapy within 2 weeks
* Concurrent immunotherapy
* Pregnant women
* Autoimmune disorder
* Severe or uncontrolled systemic disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 24 months
  Progression free survival at 6 months

SECONDARY OUTCOMES:
Objective response | 24 months
  • Objective response rate by RECIST v1.1 and iRECIST via CT scan or MRI after every 6-weeks
Overall survival | 24 months
  Overall survival at 6, 9, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sant Chawla, MD, Principal Investigator — Sarcoma Oncology Research Center; Neal Chawla, MD, Study Director — Sarcoma Oncology Research Center

IPD SHARING:
Plan to Share IPD: No
The study data will remain confidential until final publication of results.

REFERENCES:
- [Result] Chen X, Ren Z, Li C, Guo F, Zhou D, Jiang J, Chen X, Sun J, Yao C, Zheng S. Preclinical Study of Locoregional Therapy of Hepatocellular Carcinoma by Bioelectric Ablation with Microsecond Pulsed Electric Fields (musPEFs). Sci Rep. 2015 Apr 30;5:9851. doi: 10.1038/srep09851. Erratum In: Sci Rep. 2024 Aug 7;14(1):18339. doi: 10.1038/s41598-024-68637-8. PMID 25928327
- [Result] Jimenez M, Ng C, Iding J, et al. Single-Needle Delivery of Pulsed Electric Fields (PEF) Energy to Early-Stage Non- Small Cell Lung Cancer (NSCLC): Feasibility and Safety Near Sensitive Structures in the INCITE ES Study. JVIR. 2023; 34(3):S71-S72
- [Result] J. lding, P. Vanderlaan, M. Jimenez, J. Fernandez Garcia-Hierro, J. Flandes Aldeyturriaga, E. van der Heijden, C. Ng, R. Lau, M. Ludena, R. Carias, M. Cedeno, A. Moreno-Gonzalez, B. Hatton, W. Krimsky. Tertiary lymphoid structures (TLS) observed in non-small cell lung cancer (NSCLC) tumors treated with Pulsed Electric Fields. Journal for Immunotherapy of Cancer 2022;10(Suppl 2):Al-A1595